CLINICAL TRIAL: NCT07035964
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel Study on the Effects of Effera Human Lactoferrin on Gastrointestinal Permeability
Brief Title: Effects of Effera Human Lactoferrin at One Dose Compared to Placebo on Gut Permeability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helaina Inc. (Industry)
Collaborators: Biofortis Mérieux NutriSciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BIO-2504
Record Dates: First submitted 2025-06-06; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Gut Permeability; Gut Health

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement: effera human lactoferrin (Experimental): Dietary supplement: effera human lactoferrin
  Interventions: Dietary Supplement: human lactoferrin
- Dietary Supplement: Placebo Control (Placebo Comparator): Dietary Supplement: Placebo Control
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: human lactoferrin — effera human lactoferrin
  Other Names: effera
  Arms: Dietary supplement: effera human lactoferrin
Dietary Supplement: Placebo — Placebo Control
  Other Names: Control
  Arms: Dietary Supplement: Placebo Control

SUMMARY:
The purpose of this study is to evaluate the impact of 28-day supplementation with effera human lactoferrin, compared to a placebo control product on indicators of gut barrier health in males and females

DETAILED DESCRIPTION:
Samples will be retained for possible analyses such lactoferrin absorption and immune biomarkers

ELIGIBILITY:
Inclusion Criteria:

1. Male or premenopausal female, 18 - 40 years of age, inclusive
2. BMI ≥ 18.5 to < 40.0 kg/m2
3. Abdominal adiposity defined by a waist circumference >40" in men or >35" in women measured at Visit 1.
4. Reports at least mild GI symptoms from the 7d GI Symptom Questionnaire collected at visit

2. Mild GI symptoms will be defined as a combined weekly total score of gas/flatulence, abdominal distention/bloating, borborygmus/stomach rumbling, or burping symptoms ≥ 3.

5. Non-user or former user (daily use; cessation ≥ 12 months) of tobacco or nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) within 12 months of visit 1, and has no plans to begin use during the study period.

6. Non-habitual users (i.e., daily or almost daily) of marijuana or hemp products, including CBD/THC products, and willing to abstain from use throughout the study period (topical creams/lotions are allowed).

7. Willing to use personal smart phone with operating system (Android version 8.0 or newer; iOS version 15.5 or newer) capable of downloading the Cronometer app for diet records.

8. Willing to adhere to all study procedures, including lifestyle considerations ,and sign forms providing informed consent to participate in the study and authorization to release relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Clinically important GI condition that would potentially interfere with the evaluation of the study product (e.g., inflammatory bowel disease, irritable bowel syndrome, Crohn's disease, celiac disease, history of surgery for weight loss, gastroparesis, and clinically significant lactose or gluten intolerance or other food or ingredient allergies).
2. Recent (≤ 3 months of visit 1) endoscopy or colonoscopy preparation.
3. Abnormal laboratory test results of clinical significance at visit 1, at the discretion of the Clinical Investigator. One re-test will be allowed on a separate day prior to visit 2, for participants with abnormal laboratory test results.
4. Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at Visit 1. Stable use of hypertension medication is allowed (defined as no change in medication regimen within the 90 days prior to Visit 1).
5. Uncontrolled and/or clinically important pulmonary (including uncontrolled asthma), cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), hepatic, renal, endocrine (including Type 1 and Type 2 diabetes mellitus), hematologic, immunologic, neurologic (such as Alzheimer's or Parkinson's disease), psychiatric (including depression and/or anxiety disorders) or biliary disorders. Conditions that are well-controlled or resolved will be assessed by the Clinical Investigator on a case-by-case basis.
6. Unstable use (change in dose) of any prescription medications ≤ 90 d of visit 1, except for medications used PRN (e.g., asthma inhalers, non-drowsy seasonal allergy medications, etc.).
7. History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
8. Major trauma or any surgical event within 3 months of visit 1.
9. Currently scheduled, or planning to schedule, an elective surgical procedure during the study.
10. Signs or symptoms of an active infection of clinical relevance within 5 days of visit 1. The visit may be rescheduled once all signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to Visit 1. If an infection occurs during the study period, test visits will be rescheduled until signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to the scheduled study visits.
11. Diagnosis of tuberculosis of hepatitis within 1 year prior to study.
12. Extreme dietary habits (e.g., ketogenic, very high protein, very high fiber, vegan/vegetarian) at the discretion of the Clinical Investigator.
13. Weight loss or gain >4.5 kg in the 3 months prior to visit 1.
14. Currently or planning to be on a weight loss regimen during the study.
15. Recent history (≤ 12 months visit 1) of alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 11⁄2 oz distilled spirits).
16. Antibiotic use within 3 months of visit 1 and throughout the study period.
17. Recent use of oral or injectable steroids, or topical or inhaled steroids (≥ 1500 μg/d), ≤ 90 dof visit 1.
18. Regular use (≥ 3 days/week ≤ 1 month of visit 1) of anti-inflammatory medications (e.g., NSAIDS) and throughout the study period.
19. Use of medications (over-the-counter or prescription) and/or dietary supplements known to influence GI function, including but not limited to: pre-, post-, and probiotic supplements, fiber supplements, laxatives, enemas, suppositories, H2 blockers, proton pump inhibitors, antacids, anti-diarrheal agents, anti-depressants, and/or anti-spasmodic within 2 weeks of visit 1 and throughout the study period.
20. Recent use of dietary supplements containing bovine lactoferrin or iron in excess of the RDA (within 60 d of Visit 1). Standard multivitamin and mineral supplements are allowed.
21. Exposure to any non-registered drug product within 1 month of visit 1 and throughout the study period.
22. Pre-menopausal females with an irregular menstrual cycle (regular cycle defined as 21 to 35 days in length for the last 3 months prior to visit 1).
23. Female who is diagnosed with Premenstrual Dysphoric Disorder (PMDD).
24. Female who reports only experiencing GI symptoms around the time of menses.
25. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. Women who become pregnant during the study will be discontinued.
26. Female who is unwilling to adhere to medically-recognized forms of birth control (e.g., hormonal and non-hormonal contraceptives, barrier methods, abstinence, etc).
27. Female who is unwilling to wear a tampon during the collection of urine samples when these collections occur during the time of menstruation.
28. Known sensitivity, intolerability, or allergy to any of the study products, study foods, or their excipients.
29. Has a condition the Clinical Investigator believes would interfere with his ability to provide informed consent, and comply with the study protocol, which might confound the interpretation of the study results, or put the participant at undue risk.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
lactulose to mannitol ratio | 0, 4 weeks
  Change from baseline of lactulose to mannitol ratio

SECONDARY OUTCOMES:
Markers of gut barrier function | 0, 4 weeks
  Change from baseline in markers of gut barrier function (such as the change in 2-8 h urine LMR from baseline to day 28, change in 7d GI Symptom Questionnaire scores from baseline to day 28, change in Digestion-associated Quality of Life Questionnaire (DQLQ) score from baseline to day 28 and change in fasting plasma LBP concentrations from baseline to day 28)

OTHER OUTCOMES:
Questionnaire of women's health | 0, 4 weeks
  The change in (Menstrual Distress Questionnaire) MEDI-Q scores from baseline to day 28 in women participants experiencing a menses during the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis Inc, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided